CLINICAL TRIAL: NCT06867185
Title: Function And Speed of Transection Recovery After Therapeutic Electrostimulation of Nerves
Brief Title: Evaluating Therapeutic Electrical Stimulation to Improve Nerve Healing After Surgical Repair of Digital Nerve Injuries
Acronym: FASTR-TEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Checkpoint Surgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0153-CSP-300
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Digital Nerve Injury; Nerve Injury; Nerve Reconstruction; Nerve Trauma; Digital Nerve Lesion
Keywords: Nerve Repair; Therapeutic Electrical Stimulation; BES; Brief Electrical Stimulation
MeSH Terms: interventions — Electric Stimulation Therapy; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard of Care Repair (Active Comparator): Individuals will receive standard of care surgical repair of their digital nerve injury as determined by their surgeon.
  Interventions: Procedure: Digital Nerve Repair
- Repair + Therapy (Experimental): During the surgical repair for digital nerve injury (standard of care), a 10 minute dose of therapeutic electrical stimulation will be delivered during surgery.
  Interventions: Device: Brief Electrical Stimulation Therapy; Procedure: Digital Nerve Repair

INTERVENTIONS:
Device: Brief Electrical Stimulation Therapy — 10-minutes of electrical stimulation to repaired nerve
  Other Names: BES; Therapeutic Electrical Stimulation; Electrical Stimulation
  Arms: Repair + Therapy
Procedure: Digital Nerve Repair — Standard of care surgical repair of digital nerve injury as determined by health care provider.
  Other Names: Nerve Repair

SUMMARY:
The goal of this clinical study is to evaluate if a period of electrical stimulation delivered during the surgical repair procedure can speed up nerve healing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Candidate for surgical intervention under general anesthesia.
* Require primary nerve injury repair in at least 1 digital nerve.
* Following resection, have a resulting nerve gap of ≤ 10mm.
* Able to complete tension-free end-to-end direct repair, or repair with a conduit, autograft, or allograft with a length ≤15mm
* Signed and dated informed consent form.

Exclusion Criteria:

* Severe comorbid conditions, such as arrhythmia or congestive heart failure, preventing surgery under general anesthesia.
* Nerve repair occurring >1 month post-injury.
* Incomplete nerve transection.
* Injury requiring replantation of target digit
* Injury distal to the distal interphalangeal joint.
* Injury proximal to branching into the proper or common digital nerves.
* Injuries to both digital arteries of an affected digit.
* History of neuropathy, diabetic neuropathy, or any other known neuropathy
* History of chronic ischemic condition of the upper extremity
* Cognitive impairment preventing the ability to provide consent, follow post-operative instructions, or complete clinical assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Two Point Discrimination | 2 weeks - 9 months
  Evaluation of sensory function based on ability to discern two point of contact for different distances between the contacts (2-15mm). Evaluated at each follow-up visit.

SECONDARY OUTCOMES:
Semmes-Weinstein Monofilament Test | 2 weeks - 9 months
  Evaluation of sensory function, measuring pressure detection threshold. Evaluated at each follow-up visit.
Visual Analog Scale (VAS) | 2 weeks - 9 months
  Self reported rating of pain marked on a 100mm visual analog scale. Evaluated at each follow-up visit.
quick Disabilities of Arm, Hand, and Shoulder (quickDASH) | 2 weeks - 9 months
  Questionnaire providing patient reported estimate upper extremity function following injuries or disorders to the arm, hand, or shoulder. Responses to 11 questions answered on a 1-5 scale are used to calculate a scorescore ranging from 0 (no disability) to 100 (most severe disability). Evaluated at each follow-up visit.
Michigan Hand Outcomes Questionnaire (MHQ) | 2 weeks - 9 months
  A patient reported questionnaire consisting of 37 questions answered on a 1-5 scale used to calculate an estimate of hand function on a 0-100 scale with a higher number indication greater hand function. Evaluated at each follow-up visit.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - University of Missouri Department of Orthopaedic Surgery, Columbia, Missouri
  - Washington University in St Louis, Department of Orthopedic Surgery, St Louis, Missouri
  - The Ohio State Univeristy - Department of Plastic and Reconstructive Surgery, Columbus, Ohio
  - Harborview Medical Center - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Roh J, Schellhardt L, Keane GC, Hunter DA, Moore AM, Snyder-Warwick AK, Mackinnon SE, Wood MD. Short-Duration, Pulsatile, Electrical Stimulation Therapy Accelerates Axon Regeneration and Recovery following Tibial Nerve Injury and Repair in Rats. Plast Reconstr Surg. 2022 Apr 1;149(4):681e-690e. doi: 10.1097/PRS.0000000000008924. PMID 35139047
- [Background] Sayanagi J, Acevedo-Cintron JA, Pan D, Schellhardt L, Hunter DA, Snyder-Warwick AK, Mackinnon SE, Wood MD. Brief Electrical Stimulation Accelerates Axon Regeneration and Promotes Recovery Following Nerve Transection and Repair in Mice. J Bone Joint Surg Am. 2021 Oct 20;103(20):e80. doi: 10.2106/JBJS.20.01965. PMID 34668879
- [Background] Saffari TM, Walker ER, Pet MA, Moore AM. Brief Intraoperative Electrical Stimulation to Enhance Nerve Regeneration. Plast Reconstr Surg Glob Open. 2024 Apr 10;12(4):e5730. doi: 10.1097/GOX.0000000000005730. eCollection 2024 Apr. No abstract available. PMID 38600968
- [Background] Wong JN, Olson JL, Morhart MJ, Chan KM. Electrical stimulation enhances sensory recovery: a randomized controlled trial. Ann Neurol. 2015 Jun;77(6):996-1006. doi: 10.1002/ana.24397. Epub 2015 May 4. PMID 25727139